CLINICAL TRIAL: NCT02608437
Title: A Phase 1b, Open-label, Dose Escalation Study Investigating Different Doses of SGI-110 in Combination With Ipilimumab in Unresectable or Metastatic Melanoma Patients
Brief Title: A Study Investigating SGI-110 in Combination With Ipilimumab in Unresectable or Metastatic Melanoma Patients
Acronym: NIBIT-M4
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Italian Network for Tumor Biotherapy Foundation (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIBIT-M4
Record Dates: First submitted 2015-11-13; First posted 2015-11-18 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Metastatic Melanoma
Keywords: melanoma; ipilimumab; SGI-110
MeSH Terms: conditions — Melanoma | interventions — guadecitabine; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SGI-110 and Ipilimumab (Experimental): SGI-110 in combination with Ipilimumab
  Interventions: Drug: SGI-110; Drug: Ipilimumab

INTERVENTIONS:
Drug: SGI-110 — SGI-110: start at 30 mg/m2 s.c. on W0, 3, 6, 9 Day 1 - 5 q21 days. Dose level -1: 15 mg/m2; dose level +1: 45 mg/m2
Drug: Ipilimumab — ipilimumab: 3 mg/Kg i.v. over 90 minutes on W1, 4, 7 and 10 for a total of 4 cycles.
  Other Names: Ipilimumab(Yervoy)

SUMMARY:
Thi pahse I, dose-escalation trial will determine the MTD, safety and the additional benefit achieved from adding SGI-110 to ipilimumab therapy in metastatic melanoma patients. Preclinical evidence generated with SGI-110 in vivo demonstrated that besides having a direct activity on tumor growth as a single agent, SGI-110 was able to "sensitize" neoplastic cells to the anti-tumor activity of CTLA-4 blockade, providing a sound scientific rationale to develop new immunotherapeutic approaches combining SGI-110 with therapeutic mAb to immune check-points.

DETAILED DESCRIPTION:
Epigenetic alterations play a pivotal role in cancer development and progression. Pharmacologic reversion of such alterations is feasible, and second generation "epigenetic drugs" are in development and have demonstrated to possess significant immunomodulatory properties. This knowledge, together with the availability of new and highly effective immuno-therapeutic agents including immune check-point(s) blocking monoclonal antibodies, allows us to plan for highly innovative proof-of-principle combination studies that will likely open the path to more effective anti-cancer therapies.

Targeting immune check-point(s) with immunomodulatory monoclonal antibody (mAb) is a novel and rapidly evolving strategy to treat cancer, that is rapidly spreading to different tumor histologies. The prototype approach of this therapeutic modality relies on the inhibition of negative signals delivered by CTLA-4 expressed on T lymphocytes. CTLA-4 blockade has profoundly changed the therapeutic landscape of metastatic melanoma (MM), significantly improving the survival of MM patients; however, objective clinical responses are limited, and only a minority of patients achieves long-term disease control.1 Therefore, several combination approaches are being explored to improve the efficacy of CTLA-4 blockade. Along this line, based on the preclinical evidence the investigators gained on the broad immunomodulatory activity of SGI-110, the exploratory phase 1 combination study NIBIT-M4 has been designed to provide proof-of-concept evidence to the immunologic and clinical efficacy of CTLA-4 blockade combined with DNA-HypomethylatingAgent (DHA). Progressing Stage III or Stage IV MM patients, amenable to serial tumor biopsies will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* Unresectable Stage III or Stage IV melanoma with measurable lesions by CT or MRI per mWHO/irRC criteria, that can be amenable to biopsy
* Previously treated or untreated; prior therapy may include chemotherapy or targeted therapy for metastatic disease (i.e., BRAF and/or MAP-ERK kinase (MEK) inhibitor). Prior adjuvant interferon is permitted
* Subjects with Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* 4 weeks or greater since last treatment
* Must have recovered from any acute toxicity associated with prior therapy
* Life expectancy greater than 16 weeks
* Negative screening tests for HIV, Hepatitis B, and Hepatitis C
* Women of child-bearing potential must not be pregnant or breastfeeding, must have a negative pregnancy test at Screening and all men must be practicing two medically acceptable methods of birth control. Men should not father a child while receiving treatment with SGI-110 + ipilimumab, and for 2 months following completion of treatment. Men with female partners of childbearing potential should use effective contraception during this time

Exclusion Criteria:

* Subjects with any contraindications for ipilimumab
* Subjects with active brain metastases or leptomeningeal metastases
* Subjects with metastatic uveal melanoma
* Subjects with active, known or suspected autoimmune disease
* Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of treatment
* Subjects with symptomatic effusions on account of pleural, pericardial metastases of melanoma
* Prior treatment with an anti-Programmed Death receptor-1 (PD-1), anti-Programmed Death-1 ligand-1 (PD-L1), anti-PD-L2, or anti-CTLA-4 antibody
* Subjects who had major surgery or radiation therapy within 21 days of starting treatment
* Subjects who are unable to return for follow-up visits as required by this study

Other Exclusion Criteria:

* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of SGI-110 in combination with ipilimumab | the first 3 weeks of treatment
  The primary objective is to determine the MTD of SGI-110 in combination with ipilimumab in 21 day cycles in melanoma patients. Endpoints related to this objective include an evaluation of Dose Limiting Toxicity(s). The MTD evaluation will be based on the DLT evaluable population.

SECONDARY OUTCOMES:
Immune-related Disease Control Rate (irDCR) | weeks 24
  Immune-related Disease Control Rate (irDCR) is the proportion of treated subjects with an immune-related Best Overall Responce (ir-BOR) of confirmed irCR, confirmed irPR or irSD.
Immune-related Objective Response Rate (irORR) | weeks 24
  Immune-related Objective Response Rate (irORR) is the proportion of treated subjects with a irBOR of confirmed irCR or confirmed irPR.
Immune-related Time to Response (irTTR) | weeks 24
  Immune-related Time to Response (irTTR) is defined as the time from first dosing date until the measurement criteria are first met for overall response of irPR or irCR (whichever status comes first, and provided it is subsequently confirmed).
Immune-related Duration of Response (irDoR) | 2 years
  Immune-related Duration of Response (irDoR) for the subjects whose irBOR is irCR or irPR will be defined as the time between the date of response of confirmed irCR or confirmed irPR (whichever occurs first) and the date of irPD or death (whichever occurs first). The onset of a confirmed irCR or irPR is determined by the initial assessment of response, not by the confirmatory assessment. Note that if an assessment of irPR occurs before confirmation of irCR, the duration of immune-related response endpoint will not begin at the time that the irBOR of irCR is shown but rather at the earlier time-point showing irPR. For subjects who remain alive and have not progressed following response, irDoR will be censored on the date of last evaluable Tumor Assessment.
Immune-related progression free survival (irPFS) | 2 years
  Immune-related progression free survival (irPFS) per irRC will be defined as the time between the date of randomization and the date of progression per irRC or death, whichever occurs first. A subject who dies without reported progression per irRC will be considered to have progressed on the date of death. For those subjects who remain alive and have not progressed, irPFS will be censored on the date of last evaluable Tumor Assesment. For those subjects who remain alive and have no recorded post baseline Tumor Assessment, irPFS will be censored on the day of last clinical evaluation.

OTHER OUTCOMES:
Phenotypic/epigenetic profile of tumor samples and peripheral blood mononuclear cells | 2 years
  Changes in the immune phenotype/epigenetic profile of neoplastic cells and of immune cells.
humoral immune responses induced by treatment | 2 years
  Changes in the humoral and cellular immune responses induced by treatment will be investigated utilizing standardized and validated techniques.
Maximum Plasma Concentration [Cmax] of of SGI-110 and decitabine. | 24 hours
  Plasma samples will be prepared from blood drawn at the following time-points: Cycle 1, Day 1: pre-dose, 15 min, 30 min, 60 min, 90 min, 2 hr, 4 hr, 6 hr and 8 hr post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Di Giacomo, PhD,MD, Principal Investigator — Medical Oncology and Immunotherapy Unit, University Hospital of Siena
Locations (1):
- Medical Oncology and Immunotherapy Unit, University Hospital of Siena, Siena, Italy

REFERENCES:
- [Background] Maio M, Di Giacomo AM, Robert C, Eggermont AM. Update on the role of ipilimumab in melanoma and first data on new combination therapies. Curr Opin Oncol. 2013 Mar;25(2):166-72. doi: 10.1097/CCO.0b013e32835dae4f. PMID 23299197
- [Background] Covre A, Coral S, Di Giacomo AM, Taverna P, Azab M, Maio M. Epigenetics meets immune checkpoints. Semin Oncol. 2015 Jun;42(3):506-13. doi: 10.1053/j.seminoncol.2015.02.003. Epub 2015 Feb 14. PMID 25965370
- [Result] Kantarjian H, Oki Y, Garcia-Manero G, Huang X, O'Brien S, Cortes J, Faderl S, Bueso-Ramos C, Ravandi F, Estrov Z, Ferrajoli A, Wierda W, Shan J, Davis J, Giles F, Saba HI, Issa JP. Results of a randomized study of 3 schedules of low-dose decitabine in higher-risk myelodysplastic syndrome and chronic myelomonocytic leukemia. Blood. 2007 Jan 1;109(1):52-7. doi: 10.1182/blood-2006-05-021162. Epub 2006 Aug 1. PMID 16882708
- [Derived] Noviello TMR, Di Giacomo AM, Caruso FP, Covre A, Mortarini R, Scala G, Costa MC, Coral S, Fridman WH, Sautes-Fridman C, Brich S, Pruneri G, Simonetti E, Lofiego MF, Tufano R, Bedognetti D, Anichini A, Maio M, Ceccarelli M. Guadecitabine plus ipilimumab in unresectable melanoma: five-year follow-up and integrated multi-omic analysis in the phase 1b NIBIT-M4 trial. Nat Commun. 2023 Sep 22;14(1):5914. doi: 10.1038/s41467-023-40994-4. PMID 37739939
- [Derived] Amaro A, Reggiani F, Fenoglio D, Gangemi R, Tosi A, Parodi A, Banelli B, Rigo V, Mastracci L, Grillo F, Cereghetti A, Tastanova A, Ghosh A, Sallustio F, Emionite L, Daga A, Altosole T, Filaci G, Rosato A, Levesque M, Maio M, Pfeffer U, Croce M; EPigenetic Immune-oncology Consortium Airc (EPICA) consortium. Guadecitabine increases response to combined anti-CTLA-4 and anti-PD-1 treatment in mouse melanoma in vivo by controlling T-cells, myeloid derived suppressor and NK cells. J Exp Clin Cancer Res. 2023 Mar 18;42(1):67. doi: 10.1186/s13046-023-02628-x. PMID 36934257
- See also: Fondazione NIBIT — http://www.fondazionenibit.org/